CLINICAL TRIAL: NCT06940830
Title: A Low-interventional Study to Evaluate Long-term Effectiveness of Real-world Prophylactic Treatment With Efanesoctocog Alfa on Joint Health in People With Haemophilia A (ALTITUDE)
Brief Title: Long-term Study Evaluating Joint Health in People With Haemophilia A Receiving Real-world Prophylactic Treatment With Efanesoctocog Alfa
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.BIVV001-005; 2024-517812-31-00 (EU CTIS Number); U1111-1312-9668 (Registry Identifier: WHO Universal trial number (UTN))
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Joint Health; Prophylaxis; Factor VIII Deficiency; Blood coagulation disorder; Efanesoctogoc alfa; Coagulation protein disorder; ALTUVOCT; ALTUVIIIO
MeSH Terms: conditions — Hemophilia A; Blood Coagulation Disorders; Coagulation Protein Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Treatment Group (Other)
  Interventions: Drug: Efanesoctocog alfa

INTERVENTIONS:
Drug: Efanesoctocog alfa — Participant in this study must be prescribed efanesoctocog alfa prophylactic treatment per their standard of care from their physician. No drug will be provided by the Sponsor.

SUMMARY:
The rationale for this study is to further understand and describe the long-term prophylactic effectiveness of efanesoctocog alfa in preventing joint bleeds in a real-life setting.

DETAILED DESCRIPTION:
This is a retrospective-prospective, low-interventional study to evaluate the long-term effectiveness of real-world prophylaxis with efanesoctocog alfa on joint health in people with haemophilia A. Participants in the study must be prescribed efanesoctocog alfa at the discretion of their physicians within 6 months prior to, or at the time of, enrolment. The decision to initiate treatment with efanesoctocog alfa shall be made independently from the decision to include the patients in the study. A broad haemophilia A population (e.g. all severities [mild to severe], all ages, patients with comorbidities and/or concomitant use of anticoagulant/antiplatelet drugs, patients with previous inhibitors to Factor FVIII [FVIII]) will be eligible to enrol. The study will require mandatory on-site visits with joint assessments. A retrospective data collection on patients' haemophilia, medical, and surgical history will be performed, including previous haemophilia treatment and treated bleeding episodes from 12 months prior to initiating treatment with efanesoctocog alfa until enrolment.

The study will start with the enrolment visit during a patient's routine visit to the hospital, to check whether the patient fulfils all the inclusion criteria and none of the exclusion criteria. Study participants will have yearly on-site visits for 24 months or 36 months, depending on the time of enrolment in relation to study closure. Patients will be followed in the study as long as they are treated with efanesoctocog alfa prophylaxis which would be at the physicians' discretion. Patients will also need to agree to document any bleeding episodes they may have during the study in a study-specific paper diary. Joint assessment, Haemophilia Joint Health Score (HJHS), and completion of Patient-reported outcomes (PROs) will be conducted during the on-site visits. For patients included in the Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) group, ultrasound joint assessment will also be done at the yearly visits. The end of study (EoS) visit can be performed at the 24-month visit or the 36-month visit, depending on the time of enrolment.

The target is to enroll approximately 250 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with a diagnosis of haemophilia A.
2. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
3. Prescribed with efanesoctocog alfa prophylactic treatment within 6 months prior to study enrolment or at the latest at the enrolment visit, in accordance with local regulations.
4. Must have received prophylactic treatment(s) with any haemophilia product(s) for at least 12 months prior to being prescribed with efanesoctocog alfa treatment.
5. Have documented pre-study treatment data on haemophilia prophylaxis prescriptions and on treated bleeding episodes from the 12-months prior to being prescribed efanesoctocog alfa treatment and until enrolment into this study.
6. Willing to adhere to the visit schedule and to undergo mandatory study assessment (HJHS, PROs).
7. Willingness and the ability of the patient or their legally designated representative to document all bleeding episodes, including any treatments for those episodes.
8. For HEAD-US subgroup: Accept to undergo annual ultrasound assessment on the index joints (ankles, elbows, knees).

Exclusion Criteria:

1. Acquired haemophilia A and other blood clotting disorders than hereditary haemophilia A.
2. Any positive FVIII inhibitor result (defined as inhibitor titre ≥0.6 Bethesda unit [BU]/mL) from the medical records in connection to the switch to efanesoctocog alfa until the enrolment visit.
3. Enrolment in a concurrent clinical interventional study, or intake of an investigational medicinal product (IMP), including for haemophilia prophylaxis, within 3 months prior to enrolment in this study.
4. Patient not suitable for participation, whatever the reason, as judged by the Investigator, e.g., patient is not able or willing to perform the study assessments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Annualized joint bleeding rate (AjBR) over the prospective observation period. | Enrolment to Month 12, 24 and 36

SECONDARY OUTCOMES:
Annualized bleeding rate (ABR) over the prospective observation period. | Enrolment to Month 12, 24 and 36
Number of injections to control a bleeding event over the prospective observation period. | Enrolment to Month 12, 24 and 36
Total dose to control bleeding event over the prospective observation period. | Enrolment to Month 12, 24 and 36
  Cumulative amount of medication administered to effectively manage bleeding episodes.
Haemophilia Joint Health Score (HJHS) version 2.1 | Enrolment to Month 12, 24 and 36
  Change from enrolment in total and domain scores of HJHS per patient.
Target joint development on a patient and joint level over the prospective observation period. | Month 12, 24 and 36
  A target joint is defined as joints with 3 or more spontaneous bleeding episodes within a consecutive 6-month period.
Target joint resolution on a patient and joint level over the prospective observation period. | Month 12, 24 and 36
  A target joint is defined as joints with 3 or more spontaneous bleeding episodes within a consecutive 6-month period.
Target joint recurrency on a patient and joint level over the prospective observation period. | Month 12, 24 and 36
  A target joint is defined as joints with 3 or more spontaneous bleeding episodes within a consecutive 6-month period.
Annualised injection frequency over the prospective observation period. | Month 12, 24 and 36
Annualised efanesoctocog alfa consumption for prophylaxis and treatment of bleeds (excluding surgery) over the prospective observation period. | Month 12, 24 and 36
Reason(s) for any changes in prescribed frequency and/or dose of efanesoctocog alfa prophylaxis over the prospective observation period. | Enrolment to Month 12, 24 and 36
Change in ABR in the period of using efanesoctocog alfa vs prior haemophilia treatment. | Prospective period vs Retrospective period
Change in annualised injection frequency during the period on efanesoctocog alfa vs the period on prior haemophilia treatment. | Prospective period vs Retrospective period
Change in annualised consumption during the period on efanesoctocog alfa vs the period on prior haemophilia treatment. | Prospective period vs Retrospective period
Reason(s) for Switching to efanesoctocog alfa treatment. | Retrospective period (12 to 18 months prior to enrollment)
Investigator or Surgeon assessment of patient's haemostatic response on the International Society on Thrombosis and Haemostasis (ISTH) 4-point response for surgical procedures scale (Intraoperative and postoperative). | Within 96 hours following surgery
Number of injections and dose administered to maintain haemostasis during perioperative period for minor and major surgery. | Enrolment to 36 Months
Total efanesoctocog alfa consumption during perioperative period for minor/major surgery. | Enrolment to 36 Months
Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) | Enrolment to Month 12, 24 and 36
  Change from enrolment in total and domain score.
Treatment preference survey | Month 12
Patient Reported Outcome (PRO) of Pain Intensity | Enrolment to Month 12, 24 and 36
  Use of PROMIS SF v2.0 to measure change in patient-reported pain intensity from enrolment.
Patient Reported Outcome (PRO) of Pain Interference | Enrolment to Month 12, 24 and 36
  Use of PROMIS SF v2.0 to measure change in patient-reported pain interference from enrolment.
Patient Reported Outcome of 5-level EuroQol-5 dimensions [EQ-5D-5L] score | Enrolment to Month 12, 24 and 36
  Changes from enrolment of patient mobility, self-care, usual activities, pain/discomfort, anxiety/depression.
Patient Reported Outcome of youth EuroQol 5-dimensions [EQ-5D-Y] score | Enrolment to Month 12, 24 and 36
  Changes from enrolment of patient mobility, self-care, usual activities, pain/discomfort, anxiety/depression using child-appropriate wording.
Patient Reported Outcome of Parent Proxy EuroQol 5-dimensions [EQ-5D-Y:1] score | Enrolment to Month 12, 24 and 36
  Parent or caregiver's rating of the child's health outcomes based on mobility, self-care, usual activities, pain/discomfort, anxiety/depression.
Patient Reported Outcome of ACTIVLIM-Hemo. | Enrolment to Month 12, 24 and 36
  Measurement of activity limitations for patients with haemophilia (PwH).
Number of participants with occurrence of Serious Adverse Events (SAEs). | Enrolment to 36 months
Number of participants with occurrence of Adverse Events of Special Interest (AESIs). | Enrolment to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Swedish Orphan Biovitrum AB (publ)
Locations (24):
- Sobi Investigational Site, Zagreb, Croatia
- Czechia (3):
  - Sobi Investigational Site, Brno
  - Sobi Investigational Site, Ostrava
  - Sobi Investigational Site, Prague
- France (5):
  - Sobi Investigational Site, Bordeaux
  - Sobi Investigational Site, Marseille
  - Sobi Investigational Site, Nantes
  - Sobi Investigational Site, Paris
  - Sobi Investigational Site, Rennes
- Germany (5):
  - Sobi Investigational Site, Berlin
  - Sobi Investigational Site, Bonn
  - Sobi Investigational Site, Frankfurt am Main
  - Sobi Investigational Site, Hamburg
  - Sobi Investigational Site, Munich
- Sobi Investigational Site, Dublin, Ireland
- Spain (5):
  - Sobi Investigational Site, A Coruña
  - Sobi Investigational Site, Barcelona
  - Sobi Investigational Site, Málaga
  - Sobi Investigational Site, Palma de Mallorca
  - Sobi Investigational Site, Zaragoza
- United Kingdom (4):
  - Sobi Investigational Site, Birmingham
  - Sobi Investigational Site, Cardiff
  - Sobi Investigational Site, London
  - Sobi Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents. Patient level data will be anonymized and study documents, if applicable will be redacted to protect the privacy of trial participants.
URL: http://www.sobi.com/en/policies